CLINICAL TRIAL: NCT03782155
Title: Effect of Supplementation With b- Hydroxy Methyl Butyrate and Glutamine in Wound Healing Histology in Type 2 Diabetes and Controls Bloody Areas
Brief Title: Effect of Supplementation With HMB and Glutamine in Wound Healing on Bloody Areas
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Dr. Vanessa Fuchs Tarlovsky, Head of clinical nutrition, Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DI/17/111/03/014
Record Dates: First submitted 2018-10-15; First posted 2018-12-20 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Wound Healing; Diabetic
Keywords: wound healing, diabetes wound healing
MeSH Terms: interventions — Glutamine

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HMB and glutamine supplementation (Experimental): Patients with type 2 diabetes with supplementation HMB 3g, powder once a day and glutamine powder 14g once a day supplementation during 15 days.
  Interventions: Drug: glutamine supplementation; Drug: HMB
- placebo patients (Placebo Comparator): Patients with type 2 diabetes with placebo( calcium caseinate) supplementation during 15 days 17g of powder once a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: glutamine supplementation — powder 14g
  Other Names: Glutamine
  Arms: HMB and glutamine supplementation
Drug: HMB — powder 3g
  Arms: HMB and glutamine supplementation
Drug: Placebo — powder 17g
  Other Names: Calcic caseinate
  Arms: placebo patients

SUMMARY:
A randomized controlled clinical trial in two groups of supplementation with HMB and glutamine. Each group consist in 25 patients with bloody areas, one group will receive and intervention with HMB and Glutamine and the other will receive a placebo with calcium caseinate.

DETAILED DESCRIPTION:
A fundamental part of the integral management of wound healing in patients with bloody areas is nutrition, since it involves biochemical events that depend on the substrates it provides. Wound healing is a phase that demands higher needs of energy-protein than the requirement. Problem statement: Poor nutrition decreases, through specific phases, normal processes that allow the progression of wound healing. Nutrient deficiencies can have negative effects on wound healing by prolonging the inflammatory phase, decreasing fibroblast proliferation, and modifying collagen synthesis. Some amino acids are essential for the process, such as Glutamine and Hydroxymethylbutyrate.

Objective: To evaluate the effect of Glutamine and Hydroxymethylbutyrate supplementation over the cells involved in wound healing of bloody areas. Hypothesis: Glutamine and Hydroxymethylbutyrate supplementation promotes a positive effect over the cells involved in wound healing of bloody areas. Methodology: A randomized controlled clinical trial, in patients with diagnosis of bloody areas. They will be divided into two groups, the first will receive an intervention with Glutamine (14g) and Hydroxymethylbutyrate (3g) and a control group will receive a placebo with calcium caseinate (17g)

A sample of the affected tissue will be taken before and after the supplementation where histology will be analyzed.

Remains of tissue will be obteined during surgery wash for histology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bloody areas at hospital admission
* Hospital length stay around 15 days
* Medical treatment with surgical washing and negative pressure systems
* For the groups with diabetes, patients with diagnosis of type 2 diabetes with bloody areas.
* Patients that accepts and signs the informative consent.

Exclusion Criteria:

* patients with cancer or immunodeficiency
* patients with HbA1c < 12
* patients with collagen disease
* patients with allergy to intervention substances (HMB, glutamine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound healing:Number of cells per clauster in tissue sample of wound. | 15 days
  To evaluate the effect of supplementation in cellular differentiation. It will be counted and compared the number of cells per cluster in a tissue sample (lymphocytes, fibroblasts , macrophages and angiogeny) at the begining and after the supplementation.

OTHER OUTCOMES:
Bates- Jensen wound tool | 15 days
  To compared Bates- Jensen questionnaire will be applied two evaluations: first will be done before supplementation and second after finished the supplementation this scale consider physical characteristics of wound and give a punctuation 1 to 5 in each item ( size, depht, borders, necrosis, percentage of necrotic tissue , type of exudate, amount of exudate, skin color, edema, induration, granular tissue,epithelialization) according to this, items have a value that will be considered in a total punctuation of wound Punctuation 1-12 Health tissue 13- 59 regeneration 60. Degeneration
Biochemical serum values of CPR | 15 days
  To evaluate and compared the values of serum CPR, two different serum samples ( at the beginning and after finished the supplementation)
Biochemical serum values of creatinine | 15 days
  To evaluate and compared the values of serum creatinine, two different serum samples ( at the beginning and after finished the supplementation)
Biochemical serum values of procalcitonine | 15 days
  To evaluate and compared the values of serum procalcitonine, two different serum samples ( at the beginning and after finished the supplementation)
Bacterial growth per clauster in culture wound | 15 days
  It will be taken a bacterial culture of wound in two different moments ( at the beginning and after finished the supplementation) Will be counted the colony number per clauster and type of bacteria.
Type of bacterial growth in wound | 15 days
  It will be taken a bacterial culture of wound in two different moments ( at the beginning and after finished the supplementation) will be counted the kind of bacteria.
Glucemic control by glucose | 15 days
  Glucose control will be messured in serum sample (mg/dL) in two different moments: at the begining and after finished the supplementation.
Glucemic control by HbA1c | 15 days
  HbA1c(%) control will be messured in serum in two different moments: at the begining and after finished the supplementation.
Incidence of treatment- adverse events | 15 days
  Each day of supplementation will be performed a questionary about subjective syntoms( as abdominal pain, diarrhea, nausea, vomiting, constipation or others) of supplementation,

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Fuchs, PhD, Principal Investigator — Hospital General de México
Locations (1):
- Hospital General de México, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wild T, Rahbarnia A, Kellner M, Sobotka L, Eberlein T. Basics in nutrition and wound healing. Nutrition. 2010 Sep;26(9):862-6. doi: 10.1016/j.nut.2010.05.008. PMID 20692599
- [Background] Molnar JA, Vlad LG, Gumus T. Nutrition and Chronic Wounds: Improving Clinical Outcomes. Plast Reconstr Surg. 2016 Sep;138(3 Suppl):71S-81S. doi: 10.1097/PRS.0000000000002676. PMID 27556777
- [Background] Stechmiller JK. Understanding the role of nutrition and wound healing. Nutr Clin Pract. 2010 Feb;25(1):61-8. doi: 10.1177/0884533609358997. PMID 20130158
- [Background] Gundogdu RH, Temel H, Bozkirli BO, Ersoy E, Yazgan A, Yildirim Z. Mixture of Arginine, Glutamine, and beta-hydroxy-beta-methyl Butyrate Enhances the Healing of Ischemic Wounds in Rats. JPEN J Parenter Enteral Nutr. 2017 Aug;41(6):1045-1050. doi: 10.1177/0148607115625221. Epub 2016 Jan 29. PMID 26826258
- [Background] Bozkirli BO, Gundogdu RH, Ersoy E, Lortlar N, Yildirim Z, Temel H, Oduncu M, Karakaya J. Pilot Experimental Study on the Effect of Arginine, Glutamine, and beta-Hydroxy beta-Methylbutyrate on Secondary Wound Healing. JPEN J Parenter Enteral Nutr. 2015 Jul;39(5):591-7. doi: 10.1177/0148607113520433. Epub 2014 Jan 24. PMID 24463351
- [Background] Armstrong DG, Hanft JR, Driver VR, Smith AP, Lazaro-Martinez JL, Reyzelman AM, Furst GJ, Vayser DJ, Cervantes HL, Snyder RJ, Moore MF, May PE, Nelson JL, Baggs GE, Voss AC; Diabetic Foot Nutrition Study Group. Effect of oral nutritional supplementation on wound healing in diabetic foot ulcers: a prospective randomized controlled trial. Diabet Med. 2014 Sep;31(9):1069-77. doi: 10.1111/dme.12509. Epub 2014 Jun 19. PMID 24867069
- [Background] Wong A, Chew A, Wang CM, Ong L, Zhang SH, Young S. The use of a specialised amino acid mixture for pressure ulcers: a placebo-controlled trial. J Wound Care. 2014 May;23(5):259-60, 262-4, 266-9. doi: 10.12968/jowc.2014.23.5.259. PMID 24810310
- [Background] Harris C, Bates-Jensen B, Parslow N, Raizman R, Singh M, Ketchen R. Bates-Jensen wound assessment tool: pictorial guide validation project. J Wound Ostomy Continence Nurs. 2010 May-Jun;37(3):253-9. doi: 10.1097/WON.0b013e3181d73aab. PMID 20386331
- [Result] Salas-Gonzalez P, Sevilla- Gonzalez M de la L, Fuchs- Tarlovsky V. Effect of supplementation with glutamine and hydroxymethylbutirate over the cellsinvolved un wound healing. Int J Adv Res. 2018 Aug 31;6(8):100-6.
- [Result] Sipahi S, Gungor O, Gunduz M, Cilci M, Demirci MC, Tamer A. The effect of oral supplementation with a combination of beta-hydroxy-beta-methylbutyrate, arginine and glutamine on wound healing: a retrospective analysis of diabetic haemodialysis patients. BMC Nephrol. 2013 Jan 12;14:8. doi: 10.1186/1471-2369-14-8. PMID 23311725
- [Result] Rathmacher JA, Nissen S, Panton L, Clark RH, Eubanks May P, Barber AE, D'Olimpio J, Abumrad NN. Supplementation with a combination of beta-hydroxy-beta-methylbutyrate (HMB), arginine, and glutamine is safe and could improve hematological parameters. JPEN J Parenter Enteral Nutr. 2004 Mar-Apr;28(2):65-75. doi: 10.1177/014860710402800265. PMID 15080599